CLINICAL TRIAL: NCT02676934
Title: End Tidal Control of Sevoflurane
Acronym: EtCntrl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R-ETCNTRL
Record Dates: First submitted 2016-02-01; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Anesthesia of Living Donor Hepatectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Et group (Experimental): applying end tidal concentration as a control target for delivery of sevoflurane
  Interventions: Device: End tidal control module in Aisys anesthesia workstation
- FGF group (No Intervention): using Fresh gas control for sevoflurane delivery

INTERVENTIONS:
Device: End tidal control module in Aisys anesthesia workstation — THE USE OF AUTOMATED CONTROL OF END TIDAL SEVOFLURANE CONCENTRATION TO MAINTAIN ANESTHESIA DURING DONOR HEPATECTOMY
  Arms: Et group

SUMMARY:
the study compares the use of end tidal (Et) control of sevoflurane during anesthesia for living donor hepatectomy versus fresh gas (FGF) control. Et control is hypothesized to be as effective as FGF control with less cost and more operator satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* all donors scheduled for living donor hepatectomy in Mansoura liver transplant program

Exclusion Criteria:

* refusal

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
cost of sevoflurane during anesthesia | Intra-operative period

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes